CLINICAL TRIAL: NCT07296939
Title: Psychological Assessment and Treatment of Youth Emotional and Behavioral Dysregulation
Brief Title: Youth Emotional and Behavioral Treatment Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sherelle Harmon, Principal Investigator, Florida State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005777; U54CA267730 (NIH)
Record Dates: First submitted 2025-12-12; First posted 2025-12-22 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Standard evidence-based intervention based on child's primary diagnosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Participants will receive evidence-based treatment designed to address a wide range of emotional disorders.

SUMMARY:
This study aims to characterize key mechanisms underlying the development, maintenance, and treatment of severe irritability in a clinically heterogeneous sample of school-aged youth.

DETAILED DESCRIPTION:
Severe irritability in youth is associated with significant functional impairment and occurs across diagnostic categories. This study aims to characterize key mechanisms underlying the development, maintenance, and treatment of severe irritability in a clinically heterogeneous sample of school-aged youth. Participants will complete (a) a comprehensive, multimodal assessment - including diagnostic interviews, multi-informant behavioral ratings, and neurophysiological tasks - to evaluate core cognitive, behavioral, and psychosocial factors, and (b) evidence-based treatment (e.g., cognitive behavioral therapy). Repeated assessments throughout the study period will be used to evaluate study outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 4-17 years
* (a) a principal diagnosis of an anxiety or mood disorder per DSM-5 criteria, OR (b) parent report of clinically impairing irritability, emotional dysregulation, and/or disruptive behavior in youth
* Child and parent must be able to complete consent documents, assessments, and participate in treatment in English without a translator
* At least one parent must be available and willing to participant in both phases.

Exclusion Criteria:

* Gross neurological, sensory, or motor impairment
* History of seizure disorder, psychosis, or organic brain syndrome
* Conditions requiring acute intervention, e.g., active suicidality
* Non-English speaking child or parent

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impressions - Improvement Scale | Post-treatment (up to 28 weeks from baseline)
  Clinician-rated assessment of overall clinical change, with scores ranging from 1 (very much improved) to 7 (very much worse).
Affective Reactivity Index | Baseline to post-treatment (up to 28 weeks)
  Youth- and caregiver-reported measure of irritability, with total scores ranging from 0 to 12; higher scores indicate greater symptom severity.

SECONDARY OUTCOMES:
Behavior Assessment System for Children | Baseline to post-treatment (up to 28 weeks)
  Youth- and caregiver-reported measure of behavioral and emotional functioning; T-scores of 70 or higher indicate clinically significant symptoms.
Stop-Signal | Baseline to post-treatment (up to 28 weeks)
  Computerized task assessing inhibitory control in youth participants; longer stop-signal reaction times reflect slower inhibitory control.
Global-Local | Baseline to post-treatment (up to 28 weeks)
  Computerized task assessing set-shifting in youth participants; longer reaction times indicate poorer performance.
Letter Updating | Baseline to post-treatment (up to 28 weeks)
  Computerized task assessing working memory updating in youth participants; higher scores indicate better updating abilities.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States